CLINICAL TRIAL: NCT06899893
Title: Investigating the Impact of ITBS Stimulation on Various Brain Regions on the HPA Axis in Stroke Patients Using Resting-State EEG Data.
Brief Title: The Research Team Aims to Elucidate the Impact of ITBS (intermittent Theta Burst Stimulation) on the HPA Axis and Post-stroke Negative Emotions/depression by Conducting Human Experiments That Target Various Brain Regions.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Director, Department of Rehabilitation Medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shen-PJ-Ke-2025-1
Record Dates: First submitted 2025-03-10; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Post-stroke Depression
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stimulation of the cerebellar group using iTBS. (Experimental): In the trial, the group is anticipated to enroll 20 patients with post-stroke balance dysfunction for iTBS cerebellar stimulation.At the outset of enrollment (T0 phase), peripheral blood and saliva samples must be obtained to assess HPA axis-related indicators and to evaluate brain networks using TMS. Following the 15-day treatment period (T1 phase), the aforementioned blood samples will be collected once more for further testing. Furthermore, any adverse events will be documented, encompassing secondary cardiovascular events, epilepsy, and mortality outcomes.
  Interventions: Device: iTBS
- Stimulation of the Left Dorsolateral Prefrontal Cortex group using iTBS. (Experimental): In the trial, the group is anticipated to enroll 20 patients with post-stroke balance dysfunction for iTBS Left Dorsolateral Prefrontal Cortex stimulation.At the outset of enrollment (T0 phase), peripheral blood and saliva samples must be obtained to assess HPA axis-related indicators and to evaluate brain networks using TMS. Following the 15-day treatment period (T1 phase), the aforementioned blood samples will be collected once more for further testing. Furthermore, any adverse events will be documented, encompassing secondary cardiovascular events, epilepsy, and mortality outcomes.
  Interventions: Device: iTBS
- Stimulation of the Primary Motor Cortex (M1) group using iTBS. (Experimental): In the trial, the group is anticipated to enroll 20 patients with post-stroke balance dysfunction for iTBS Primary Motor Cortex stimulation.At the outset of enrollment (T0 phase), peripheral blood and saliva samples must be obtained to assess HPA axis-related indicators and to evaluate brain networks using TMS. Following the 15-day treatment period (T1 phase), the aforementioned blood samples will be collected once more for further testing. Furthermore, any adverse events will be documented, encompassing secondary cardiovascular events, epilepsy, and mortality outcomes.
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — Sixty patients experiencing post-stroke negative emotions were recruited and categorized into groups based on their conditions. The group with post-stroke balance dysfunction underwent intermittent theta burst stimulation (iTBS) of the cerebellum, while the group with post-stroke cognitive dysfunction received iTBS stimulation of the left dorsolateral prefrontal cortex (DLPFC), and the group with post-stroke motor dysfunction underwent iTBS stimulation of the primary motor cortex (M1).The TMS stimulation protocol consisted of 20-minute sessions, five times a week, for a total of ten sessions, utilizing a figure-of-eight coil (model B9076, coil diameter 92 mm, manufactured by Yiruide Company in Wuhan, China, transcranial magnetic therapy device model NS5000). The stimulation intensity was set at 80% of the active motor threshold, with the coil positioned tangentially to the scalp and the handle oriented upwards.

SUMMARY:
The project team will categorize stroke patients into three groups receiving iTBS stimulation targeting distinct brain regions: the cerebellum, the dorsolateral prefrontal cortex (DLPFC), and the primary motor cortex (M1), with 20 patients allocated to each group. Neurofunctional scores, anxiety and depression assessments, and transcranial magnetic stimulation evoked potentials (TEP) will be assessed pre- and post-treatment within each group. The relationship between anxiety and depression scores and brain network characteristics associated with emotions will be examined to investigate the impact of iTBS stimulation on post-stroke negative emotions. Furthermore, plasma and saliva samples will be collected from stroke patients in each group post iTBS intervention. ELISA will quantify ACTH levels in plasma and cortisol levels in both plasma and saliva, with the aim of exploring the effects of iTBS stimulation on the HPA axis across different brain regions.

ELIGIBILITY:
Inclusion Criteria:

1. Initial stroke onset <6 months, or the last stroke event occurred more than 6 months ago;
2. Age ≥18 years, <85 years (the likelihood of VCI increases beyond 85 years);
3. Patients with lesions in the middle cerebral artery region;
4. NIHSS >4, NIHSS <26;
5. mRS score ≥2;
6. Completion of CT or MRI;
7. No severe neurological or psychiatric disorders; no impairment of consciousness, able to cooperate with relevant treatments; no severe cognitive impairment (MMSE ≥15);
8. All participants are right-handed;
9. Signed informed consent form.

Exclusion Criteria:

1. History of epilepsy or psychiatric disorders (including depression, anxiety, or schizophrenia);
2. Severe comorbidities;
3. History of medication use: benzodiazepines, baclofen, or antidepressants;
4. Non-compliance with the protocol;
5. Acute phase of cerebral hemorrhage or acute infectious diseases;
6. Severe suicidal tendencies in patients with depression;
7. Severe headache, hypertension, malignant tumors, open wounds, vascular embolism, leukopenia, or other serious conditions;
8. Severe alcohol abuse;
9. History of cranial surgery or presence of metal implants in the brain;
10. Patients with cardiac pacemakers;
11. NIHSS > 26 or MMSE < 15;
12. Any condition likely to result in the patient's survival for less than 1 month;
13. Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Salivary Cortisol | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  Saliva samples were collected from stroke patients in each group post-iTBS intervention. These samples were analyzed using ELISA to quantify cortisol levels in saliva. The aim was to explore the impact of iTBS stimulation on various brain regions on the HPA axis. The concentration of cortisol in saliva is measured in nanograms per milliliter (ng/mL).
Plasma adrenocorticotropic hormone | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  Plasma samples were collected from stroke patients in each group post-iTBS intervention. These samples were analyzed using ELISA to quantify ACTH levels in plasma. The aim was to explore the impact of iTBS stimulation on various brain regions on the HPA axis. The concentration of ACTH in plasma is measured in picograms per milliliter (pg/mL).
Plasma cortisol | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  Plasma samples were collected from stroke patients in each group post-iTBS intervention. These samples were analyzed using ELISA to quantify cortisol levels in plasma. The aim was to explore the impact of iTBS stimulation on various brain regions on the HPA axis. The concentration of cortisol in plasma is measured in nanograms per milliliter (ng/mL).

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The NIHSS ranges from 0 (no stroke symptoms) to 42 (most severe stroke), with higher scores indicating worse outcomes and lower scores indicating better outcomes.
The Modified Rankin Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The Modified Rankin Scale (mRS) ranges from 0 (no symptoms) to 6 (death), with higher scores indicating worse outcomes.
Hamilton Anxiety Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The Hamilton Anxiety Scale (HAM-A) ranges from 0 (no anxiety) to 56 (severe anxiety), with higher scores indicating worse outcomes.
Hamilton Depression Rating Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The Hamilton Depression Rating Scale (HDRS) ranges from 0 (no depression) to 52 (severe depression), with higher scores indicating worse outcomes.
Self-Rating Depression Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The Self-Rating Depression Scale (SDS) ranges from 20 (no depression) to 80 (severe depression), with higher scores indicating worse outcomes.
Self-Rating Anxiety Scale | From the patient's first treatment to the completion of the 14-day iTBS therapy.
  The Self-Rating Anxiety Scale (SAS) ranges from 20 (no anxiety) to 80 (severe anxiety), with higher scores indicating worse outcomes.

IPD SHARING:
Plan to Share IPD: No